CLINICAL TRIAL: NCT02880631
Title: BAROSTIM THERAPY™ In Resistant Hypertension: A Post-Market Registry With the CE-Marked BAROSTIM NEO™ System
Brief Title: BAROSTIM THERAPY™ In Resistant Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 360051-001
Record Dates: First submitted 2016-08-15; First posted 2016-08-26 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: BAROSTIM NEO™ System

SUMMARY:
The purpose of this registry (NCT02880631) is to evaluate the effect of BAROSTIM THERAPY with the BAROSTIM NEO System in the commercial setting in subjects recently implanted under the CE-Marked indication for resistant hypertension.

DETAILED DESCRIPTION:
Summary:

The CVRx BAROSTIM THERAPY in Resistant Hypertension Registry will be performed with subjects who have been recently implanted with the BAROSTIM NEO System in accordance with CE-Mark approved criteria for resistant hypertension. Subjects must be enrolled within 30 days from implant. Up to 500 subjects will be enrolled at up to 50 sites. Data should be obtained from standard of care measurements taken prior to implant, at enrollment/baseline, and at 3, 6, and 12 months after the device was implanted. After 12 months, data may be obtained in six month intervals for up to three years after implant, at which time each subject will be exited from the registry.

Eligibility:

Subjects must sign an Ethics Committee (EC) approved informed consent form for the registry to participate.

Subjects can be included in the Hypertension Registry if they were implanted in the past 30 days and meet the CE-Mark approved indications and contraindications for the BAROSTIM NEO System in the treatment of resistant hypertension. These include:

* Indications

  * Systolic blood pressure greater than or equal to 140 mmHg, and
  * Resistance to maximally tolerated therapy with a diuretic and two other anti-hypertension medications
* Contraindications

  * Bilateral carotid bifurcations located above the level of the mandible
  * Baroreflex failure or autonomic neuropathy
  * Uncontrolled, symptomatic cardiac bradyarrhythmias
  * Carotid atherosclerosis that is determined by ultrasound or angiographic evaluation to be greater than 50%
  * Ulcerative plaques in the carotid artery as determined by ultrasound or angiographic evaluation

ELIGIBILITY:
Inclusion Criteria:

* Has signed an EC approved informed consent form
* Has been implanted with the BAROSTIM NEO system in the past 30 days
* Systolic blood pressure greater than or equal to 140 mmHg, and
* Resistance to maximally tolerated therapy with a diuretic and two other anti-hypertension medications

Exclusion Criteria:

* Bilateral carotid bifurcations located above the level of the mandible
* Baroreflex failure or autonomic neuropathy
* Uncontrolled, symptomatic cardiac bradyarrhythmias
* Carotid atherosclerosis that is determined by ultrasound or angiographic evaluation to be greater than 50%
* Ulcerative plaques in the carotid artery as determined by ultrasound or angiographic evaluation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects can be included in the Hypertension Registry if they were implanted in the past 30 days and meet the CE-Mark approved indications and contraindications for the BAROSTIM NEO System in the treatment of resistant hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-12-13 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Changes | Pre-implant baseline to 3 years post-implant
  The results of an office cuff blood pressure measurement to be obtained from a time point prior to implant and as close to the implant procedure as possible (baseline), at 3- and 6- and 12-months post-implant, and then every 6 months up to 3 years from implant.
Cardiovascular Medication Changes | Post-implant enrollment to 3 years post-implant
  Information on currently-utilized doses of cardiovascular medications will be collected at pre-implant baseline, 3- and 6- and 12-months post-implant, and then every 6 months up to 3 years from implant.
Number of Health Care Utilizations | 3 months post-implant to 3 years post-implant
  Health care utilization information (e.g. heart failure hospitalizations) is collected at 3- and 6- and 12-months post-implant, and then every 6 months up to 3 years from implant.

CONTACTS AND LOCATIONS:
Overall Officials: Hannes Reuter, PhD, Study Chair — Herzzentrum Uniklinik Köln
Locations (26):
- Germany (25):
  - Charité Benjamin Franklin, Berlin
  - Charité Campus Virchow, Berlin
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau
  - Cloppenburg Katholische Kliniken Münsterland, Cloppenburg
  - Universitätsklinikum Köln Herzzentrum, Cologne
  - Lippe Klinikum, Detmold
  - Herzzentrum Dresden, Dresden
  - Krankenhaus Erding, Erding
  - Cardiovascular Center 'CVC' Frankfurt, Frankfurt
  - Universitätsklinikum Gießen und Marburg, Giessen
  - Herzzentrum Göttingen, Göttingen
  - Asklepios Klinik Altona, Hamburg
  - St. Barbara Klinik Hamm, Hamm
  - Kardiologie im Klinikum Ingolstadt, Ingolstadt
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Herzentrum Lahr, Lahr
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinik Mainz, Mainz
  - Papenburg Marien Krankenhaus, Papenburg
  - Universitätsklinikum Regensburg, Regensburg
  - Marienkrankenhaus Siegen, Siegen
  - Krankenhaus & MVZ Maria-Hilf Stadtlohn GmbH, Stadtlohn
  - Klinikum Stuttgart, Stuttgart
  - Klinikum Tuttlingen, Tuttlingen
  - Heinrich-Braun Klinikum, Zwickau
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scheffers IJ, Kroon AA, Schmidli J, Jordan J, Tordoir JJ, Mohaupt MG, Luft FC, Haller H, Menne J, Engeli S, Ceral J, Eckert S, Erglis A, Narkiewicz K, Philipp T, de Leeuw PW. Novel baroreflex activation therapy in resistant hypertension: results of a European multi-center feasibility study. J Am Coll Cardiol. 2010 Oct 5;56(15):1254-8. doi: 10.1016/j.jacc.2010.03.089. PMID 20883933
- [Background] Bisognano JD, Bakris G, Nadim MK, Sanchez L, Kroon AA, Schafer J, de Leeuw PW, Sica DA. Baroreflex activation therapy lowers blood pressure in patients with resistant hypertension: results from the double-blind, randomized, placebo-controlled rheos pivotal trial. J Am Coll Cardiol. 2011 Aug 9;58(7):765-73. doi: 10.1016/j.jacc.2011.06.008. PMID 21816315
- [Background] Bakris GL, Nadim MK, Haller H, Lovett EG, Schafer JE, Bisognano JD. Baroreflex activation therapy provides durable benefit in patients with resistant hypertension: results of long-term follow-up in the Rheos Pivotal Trial. J Am Soc Hypertens. 2012 Mar-Apr;6(2):152-8. doi: 10.1016/j.jash.2012.01.003. Epub 2012 Feb 15. PMID 22341199
- [Background] Hoppe UC, Brandt MC, Wachter R, Beige J, Rump LC, Kroon AA, Cates AW, Lovett EG, Haller H. Minimally invasive system for baroreflex activation therapy chronically lowers blood pressure with pacemaker-like safety profile: results from the Barostim neo trial. J Am Soc Hypertens. 2012 Jul-Aug;6(4):270-6. doi: 10.1016/j.jash.2012.04.004. Epub 2012 Jun 12. PMID 22694986
- See also: BAROSTIM THERAPY website — https://www.barostimtherapy.com/